CLINICAL TRIAL: NCT01598974
Title: Brain Plasticity Underlying Back Pain Response to Different Acupuncture Methods
Brief Title: Back Pain Response to Different Acupuncture Methods
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Robert Edwards, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011P001364
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Lower Back Pain
Keywords: Lower Back Pain; Acupuncture
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Traditional Acupuncture (Experimental): Participants will receive acupuncture over 6 30-minute sessions.
  Interventions: Procedure: Traditional Acupuncture
- Laser Acupuncture (Experimental): Participants will receive laser acupuncture over 6 30-minute sessions.
  Interventions: Procedure: Laser Acupuncture
- Wait-List (No Intervention): Subjects will be put on a 6 week wait-list and receive vouchers for acupuncture at a local clinic.

INTERVENTIONS:
Procedure: Traditional Acupuncture
  Arms: Traditional Acupuncture
Procedure: Laser Acupuncture
  Arms: Laser Acupuncture

SUMMARY:
Acupuncture has been used for many years to help relieve pain. However, it is not clear how acupuncture works. We are doing this study to learn about the effects of different forms of acupuncture on chronic low back pain. We are interested in learning about brain activity during pain. We plan to look at brain activity at the beginning and the end of the study, after 6 sessions of acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers 18-60 years of age.
* Meet the Classification Criteria of the chronic LBP (having low back pain for more than 6 months), as determined by the referring physician.
* At least 4/10 clinical pain on the 11-point LBP intensity scale.
* Patients must be able to provoke or exacerbate their chronic LBP using our calibrated exercise-like maneuver.
* Must have had a prior evaluation of their low back pain by a health care provider, which may have included radiographic studies. Documentation of this evaluation will be sought from Partners or outside medical records and kept in the subject's research record.
* At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Specific causes of back pain (e.g. cancer, fractures, spinal stenosis, infections),
* Complicated back problems (e.g. prior back surgery, medicolegal issues),
* Possible contraindications for acupuncture (e.g. coagulation disorders, cardiac pacemakers, pregnancy, seizure disorder), and conditions that might confound acupuncture intervention effects or interpretation of results (e.g. severe fibromyalgia, rheumatoid arthritis).
* Conditions making acupuncture difficult (e.g. paralysis, psychoses),
* Prior acupuncture treatment for back pain; 1 year wait for any other type.
* The intent to undergo surgery during the time of involvement in the study.
* History of cardiac, respiratory, or nervous system disease that, in Dr. Wasan's judgment, precludes participation in the study because of a heightened potential for adverse outcome. For example: asthma or claustrophobia.
* Presence of any contraindications to MRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy.
* Involvement in workmen's compensation or disability claims.
* Radicular pain extending below the knee.
* Active substance abuse disorders within the last 24 months, based on subject self-report.
* Use of more than 60 mg morphine equivalent prescription opioids or steroids for pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Pain improvement in patients with lower back pain | 6 weeks
  Pain rating changes for chronic low back pain after acupuncture sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Edwards, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- MGH - Martinos Center, Charlestown, Massachusetts, United States